CLINICAL TRIAL: NCT06871384
Title: Polyphenols From Nonalcoholic Red Wine and Healthy Aging: an Opportunity to Understand Diet Modulation of the Aging Process From a Multidimensional Perspective
Brief Title: Dietary Strategy to Tackle Cognitive and Locomotor Abilities in Early Elderly Subjects
Acronym: WinAging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Rosa Sola, Full Professor, Dr. Rosa Solà Alberich, University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WinAging Study; PID2023-148704OB-C22 (Other Grant/Funding Number: The present study is funded by MICIU/AEI/10.13039/501100011033 and by FEDER, UE)
Record Dates: First submitted 2025-02-21; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Disorders; Muscular Disorders, Atrophic
Keywords: cognitive impairment; locomotor impairment; sarcopenia; aging; mediterrnean diet; non-alcoholic wine; polyphenols
MeSH Terms: conditions — Cognitive Dysfunction; Muscular Disorders, Atrophic; Sarcopenia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized, controlled parallel intervention study. The total duration of the intervention will be 9 months. Subjects will be assigned to participate in any of the two groups in a randomized fashion:
  1. Intervention group: Mediteranean diet + nonalcoholic red wine (300 mL wine/day, equivalent to a daily dose of 150 mg red wine polyphenols/day, during meals)
  2. Control group (Group B): Mediterranean diet + drinking water (300 mL/day, during meals).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nonalcoholic red wine group (Intervention group) (Experimental): Mediteranean diet + nonalcoholic red wine
  Interventions: Dietary Supplement: Nonalcoholic red wine group (Intervention group)
- Drinking water group (Control group) (Placebo Comparator): Mediterranean diet + drinking water
  Interventions: Dietary Supplement: Drinking water group (Control group)

INTERVENTIONS:
Dietary Supplement: Nonalcoholic red wine group (Intervention group) — Mediteranean diet + nonalcoholic red wine (300 mL wine/day, equivalent to a daily dose of 150 mg red wine polyphenols/day, during meals)
  Arms: Nonalcoholic red wine group (Intervention group)
Dietary Supplement: Drinking water group (Control group) — Mediterranean diet + drinking water (300 mL/day, during meals)
  Arms: Drinking water group (Control group)

SUMMARY:
Polyphenols, precisely resveratrol, with red wine as the most substantial source, was associated with improvements in cognitive function. Also, the loss of muscle mass and strength in elderly, that significantly increases dependency of these people, it could be attributed to alterations in gut microbiota through the "gut-muscle axis" and this underline the urgent need to efficiently find out any intervention or preventive approach via modulation of gut microbiota to improve muscle function in elderly. In this context, red wine polyphenols exert their effects through interaction with gut microbiota following the well-known two-way interaction between polyphenols and gut microbiota by promoting the proliferation of beneficial bacteria and increasing their abundance. Similarly, aging cognitive decline can be modulate by microbiota, notably through "gut-brain axis". Additionally, dietary polyphenols can delay inflammation or/and oxidation on the onset of age-related cognitive decline or muscular oxidation or cardiovascular factors risk factors, all of them relevant factors for the onset of physical frailty and dependence in elderly.

Moreover, wine is a singular alcoholic beverage with a high content of phenolic compounds of a very diverse nature on which numerous protective effects on health have been described. In fact, wine, in addition to alcohol, contains a complex mixture of polyphenols, including anthocyanins and non-coloured phenols as proanthocyanidins, flavonols, hydroxycinnamic and hydroxybenzoic acids, stilbenes and lignans. Thus, the bioprotective effects of wine polyphenols could be the consequence of the synergistic effect of this complex mixture of polyphenols from the grape and the winemaking process. That is why it is essential to clarify whether consumption of polyphenols from red wine provided by a nonalcohol red wine within a healthy diet can produce beneficial effects on health, differentiating this pattern from a general consumption of alcohol generally associated with negative effects. Based on the ethical limitations to carry out diet intervention studies with wine in humans, this project proposes the use of a nonalcoholic wine as vehicle of the complex mixture of red wine polyphenols.

The hypothesis of our research is that regular consumption of red wine polyphenols, 150 mg/day, delivered through a nonalcoholic red wine, in the context of a Mediterranean diet (MD pattern), could promote protective mechanisms for a healthy aging, especially through its beneficial effects on cognitive and locomotor abilities and mediated by the modulation of the intestinal microbiota (composition, function and associated metabolome). The main objective of the WinAging project is to add knowledge concerning the diet modulation of molecular mechanisms of the aging process through multi-omic approaches based on the potential health effects of a dietary strategy by a sustained MD supplementation with nonalcoholic red wine rich in polyphenols to tackle cognitive and locomotor abilities in early elderly home-dwelling subjects.

The specific objectives:

* Objective 1. To develop a nonalcoholic red wine with high phenolic content and sensorial acceptability.
* Objective 2. To evaluate the chronic effects of the intake of wine polyphenols (average dose 150 mg/day) delivered through a nonalcoholic red wine in the context of a MD in early elderly home-dwelling subjects, and applying participatory research to increase adherence of subjects in the clinical intervention study.

  * Objective 2.1. To identify selective biological phenolic metabolites in human urine samples to be used as biomarkers of nonalcoholic red wine intake.
  * Objective 2.2. To assess the effects of the diet supplementation with red wine polyphenols on the improvement of cognitive ability.
  * Objective 2.3. To assess the effects of the diet supplementation with red wine polyphenols on the improvement of locomotor ability
  * Objective 2.4. To evaluate the effect of the diet supplementation with red wine polyphenols on the improvement of cardiovascular disease (CVD) risk factors.
* Objective 3. To unravel the underlying mechanisms involved in the potential beneficial effects of red wine polyphenols on aging.

  * Objective 3.1. To evaluate the influence on microbiota composition, function and microbial catabolites.
  * Objective 3.2. To evaluate the impact on inflammation and gut health.
  * Objective 3.3. To evaluate the impact on metabolic pathways related with aging
  * Objective 3.4. To analyze the impact on age-related epigenetic modifications
  * Objective 3.5. To deeply characterize the underlying muscle signalling pathways affected using an animal model of aging.
* Objective 4. To apply integrative computational analyses for the identification of variables (clinical or gut-related) more determinant for a successful prevention of locomotor and cognitive abilities associated with wine polyphenols.

DETAILED DESCRIPTION:
A total of 72 home-dwelling early elderly volunteers (men and women) 60-74 years old will be included in the intervention (36 in each arm of the intervention).

During the study there will be 11 visits in total. Visits will be every 4 weeks form the V1. The study visits will be the following:

* Screening visit (V0).
* Basal visit (V1).
* Visits during intervention (V2, V3, V4, V5, V6, V7, V8, V9).
* 3-month study visit (V4)
* 6-month study visit (V7)
* Telephone visits (V2, V3, V5, V6, V8, V9)
* Final study visit (V10). In visits V0, V1, V4, V7 and V10 volunteers must present themselves in fasting conditions of 8 hours to obtain fasting blood samples.

  * In addition, future candidates will be provided with the nonalcoholic wine, selected for study and allowed to taste it for one week to check its tolerability and sensory acceptance and thus ensure that candidates can commit to drinking the study wine daily for 9 months and reduce follow-up losses during the intervention.

Basal visit (V1; week 0):

* Nuclear Magnetic Resonance (NMR) and muscle biopsy (±5 days V1)*.
* Isokinetic assessment (±5 days V1)*
* Revision of study clinical history.
* Vital signs (blood pressure/resting heart rate).
* Checking the concomitant medication.
* Anthropometry waist circumference; hip; body weight and composition; height).
* Checking the physical activity and sedentary habits (IPAQ-E).
* Checking the quality of life (SF-36 Health survey questionnaire)
* Checking depression symptoms (Geriatric Depression Scale Questionnaire)
* Checking MD adherence
* Checking the cognitive and locomotor abilities
* Spanish validated of the Mini Mental State Examination (MMSE), Alzheimer disease questionnaire (AD8), Memorey Alteration tets (TAM test), Fototest
* Sarcopenic parameters (muscle strength based on grip dynamometry; skeletal muscle mass index (SMI) based on bioimpedance analysis (BIA), kg/m2 and appendicular skeletal muscle mass index (ASMI) based on bioimpedance analysis (BIA), low physical performance or physical function based on 4 m gait speed, m/s.
* Blood sample extraction.
* Ultrasound (muscle mass and abdominal fat).
* Checking the 3-day dietary record and Food Frequency Questionnaire (FFQ).
* Collection of feaces samples.
* Collection of saliva samples.
* Collection of urine samples.
* MD guidelines explanation.
* Schedule the next visit and instructions.
* Administration of red nonalcoholic wine through opaque bottles to protect from light.

  * In a subsample of n= 15 subjects/group, 5 days before or after the visit V1, volunteers must have a:

    * NMR, in order to measure changes in hippocampal volume, and volume of white matter hyperintense lesions,
    * Muscle biopsys, in order to measure changes in signalling pathways in skeletal muscle,
    * Isokinetics analysis in order to measure changes in muscle function through variables such as torque, work and power.

Telephone visits: (V2 and V3; week 4 and 8):

* Checking the FFQ
* Checking changes in concomitant medication
* Product intake control
* Record adverse effects
* Schedule the next visit and instructions.

  3-month study visit (V4; week 12):
  * Revision of study clinical history.
  * Vital signs (blood pressure/resting heart rate).
  * Checking the concomitant medication.
  * Anthropometry waist circumference; hip; body weight and composition; height).
  * Checking the physical activity and sedentary habits (IPAQ-E).
  * Checking the quality of life (SF-36 Health survey questionnaire)
  * Checking depression symptoms (Geriatric Depression Scale Questionnaire)
  * Checking MD adherence
  * Checking the cognitive and locomotor abilities
  * Spanish validated of the MMSE, AD8, TAM test, Fototest
  * Sarcopenic parameters (muscle strength based on grip dynamometry; skeletal muscle mass index (SMI) based on bioimpedance analysis (BIA), kg/m2 and appendicular skeletal muscle mass index (ASMI) based on bioimpedance analysis (BIA), kg/m2; low physical performance or physical function based on 4 m gait speed, m/s.
  * Blood sample extraction.
  * Ultrasound (quadricep muscle mass and abdominal fat).
  * Checking the Food Frequency Questionnaire, Mediterranean adherence (FFQ).
  * Collection of urine samples.
  * Product intake control
  * Record adverse effects
  * MD guidelines explanation.
  * Schedule the next visit and instructions.
  * Administration of red nonalcoholic wine through opaque bottles to protect from light.

Telephone visits: (V5 and V6; week 16 and 20):

* Checking the FFQ
* Checking changes in concomitant medication
* Product intake control
* Record adverse effects
* Schedule the next visit and instructions. 6-month study visit (V7; week 24):

  * Revision of study clinical history.
  * Vital signs (blood pressure/resting heart rate).
  * Checking the concomitant medication.
  * Anthropometry waist circumference; hip; body weight and composition; height).
  * Checking the physical activity and sedentary habits (IPAQ-E).
  * Checking the quality of life (SF-36 Health survey questionnaire)
  * Checking depression symptoms (Geriatric Depression Scale Questionnaire)
  * Checking MD adherence
  * Checking the cognitive and locomotor abilities
  * Spanish validated of the MMSE, AD8, TAM test, Fototest
  * Sarcopenic parameters (muscle strength based on grip dynamometry; skeletal muscle mass index (SMI) based on bioimpedance analysis (BIA), kg/m2 and appendicular skeletal muscle mass index (ASMI) based on bioimpedance analysis (BIA), kg/m2; low physical performance or physical function based on 4 m gait speed, m/s.
  * Blood sample extraction.
  * Ultrasound (quadricep muscle mass and abdominal fat).
  * Checking the 3-day dietary record and Food Frequency Questionnaire (FFQ).
  * Collection of feaces samples.
  * Collection of saliva samples.
  * Collection of urine samples.
  * MD guidelines explanation.
  * Schedule the next visit and instructions.
  * Administration of red nonalcoholic wine through opaque bottles to protect from light.

Telephone visits: (V8 and V9; week 28, and 32):

* Checking the FFQ
* Checking changes in concomitant medication
* Product intake control
* Record adverse effects
* Schedule the next visit and instructions.

Final visit (V10; week 36):

* NMR and muscle biopsy (±5 days V1)*.
* Isokinetic assessment (±5 days V1)*
* Revision of study clinical history.
* Vital signs (blood pressure/resting heart rate).
* Checking the concomitant medication.
* Anthropometry waist circumference; hip; body weight and composition; height).
* Checking the physical activity and sedentary habits (IPAQ-E).
* Checking the quality of life (SF-36 Health survey questionnaire)
* Checking depression symptoms (Geriatric Depression Scale Questionnaire)
* Checking MD adherence
* Checking the cognitive and locomotor abilities
* Spanish validated of the MMSE, AD8, TAM test, Fototest
* Sarcopenic parameters (muscle strength based on grip dynamometry; skeletal muscle mass index (SMI) based on bioimpedance analysis (BIA), kg/m2 and appendicular skeletal muscle mass index (ASMI) based on bioimpedance analysis (BIA), kg/m2; low physical performance or physical function based on 4 m gait speed, m/s.
* Blood sample extraction.
* Ultrasound (quadricep muscle mass and abdominal fat).
* Checking the 3-day dietary record and Food Frequency Questionnaire (FFQ).
* Collection of feaces samples.
* Collection of saliva samples.
* Collection of urine samples. *In a subsample of n= 15 subjects/group, 5 days before or after the visit V10.

  * Nuclear Magnetic Resonance (NMR), in order to measure changes in hippocampal volume, and volume of white matter hyperintense lesions,
  * Muscle biopsys, in order to measure changes in signalling pathways in skeletal muscle,
  * Isokinetics analysis in order to measure changes in muscle function through variables such as torque, work and power.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between 60-74 years old; Sensory tolerance to red wine; Written informed consent provided before the initial screening visit.

Exclusion Criteria:

1. Men or women >75 years old,
2. Hypoglucaemiant treatment or type 1 and type 2 diabetes mellitus diagnosed
3. Anaemia (hemoglobin ≤13 g/dL in men and ≤12 g/dL in women)
4. Subjects diagnosed of intestinal disorders such as chron disease, colitis ulcerous, and irritable bowel syndrome
5. To present a clinical active chronic disease
6. To present severe sarcopenia
7. To present cognitive impairment (MMSE ≤ 24 or clinical diagnosis of mild cognitive impairment or dementia)
8. Dietary allergies to: Mediterranean foods (eg, nuts), sulphytes or nitrates
9. Use of antioxidants supplements
10. Regular consumers of red wine who do not agree to change the consumption of red wine with alcohol to nonalcholized wine during the intervention
11. Chronic alcoholism
12. Current or past participation in a clinical trial or consumption of a research product in the 30 days prior to inclusion in the study
13. Failure to follow the study guidelines. For participation in the muscle biopsy, additional exclusion criteria included: Use of prescription anti-platelet medication; Prescription anticoagulant use (or antiaggregant, or acenocoumarol; Conditions which would reduce healing; or known allergy to lidocaine.

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | Visit 0 (week -1), visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  The MMSE test for cognitive function. The total test score ranges from 0 (impaired) to 30 (normal) (Beaman et al., 2004).
Muscle strength | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  The muscle strength based on handgrip dynamometry (Jamar dynamometer; Sammons Preston Rolyan, Bolingbrook, IL)

SECONDARY OUTCOMES:
Anthropometric measures | Visit 0 (week -1), visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  WC: waist circumference (cm) measured by steel measuring tape (at the umbilicus)
Anthropometric measures | Visit 0 (week -1), visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Height (cm) measured by wall-mounted stadiometer (Tanita Leicester Portable; Tanita Corp., Barcelona, Spain)
Anthropometric measures | Visit 0 (week -1), visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Weight (kg) measured by calibrated scale (TANITA MC-780MA; Tanita Corp., Tokyo, Japan).
Anthropometric measures | Visit 0 (week -1), visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  BMI (kg/m2) calculated by weight (kg) divided to height (m2).
Anthropometric measures | Visit 0 (week -1), visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Body composition (Fat mass (% and kg)) measured by calibrated scale (TANITA MC-780MA; Tanita Corp., Tokyo, Japan).
Physical activity compliance | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  International physical activity questionnaire for elderly: IPAQ for elderly IPAQ-E Spanish version (Rubio-Castañeda et al., 2017). Higher scores mean a better outcome.
Sedentary habits | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Questionnaire developed by Marshall et al 2010. Higher amount of hours mean bad outcome.
Sleep quality | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Pittsburgh questionnaire (Buysse et al., 1989). The maximum score is 21 points. More than 5 points are considered bad outcomes and sleep problems, and less than 5 points are considered better outcomes and no sleep problems.
Life quality | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  SF-36 Health survey questionnaire (Ware & Sherbourne, 1992). Higher scores mean a better outcome.
Depressive symptoms | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Geriatric Depression Scale Questionnaire (Yesavage et al., 1983). The maximum puntuation is 15. The score is 0-4 no depression, 5-8 mild depression, 9-11 moderate depression and 12-15 severe depression.
Nutritional intake | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  3-day dietary record
Nutritional intake | Visit 1 (week 0), visit 2 (week 4), visit 3 (week 8), visit 4 (week 12), visit 5 (week 16), visit 6 (week 20), visit 7 (week 24), visit 8 (week 28), visit 9 (week 32), visit 10 (week 36))
  FFQ MD adherence to assess food groups intake (Martinez-Gonzalez et al., 2012) Higher scores mean a better outcome.
Nutritional status | Visit 0 (week -1)
  Mini Nutrition Assessment (MNA)
Nutritional status | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Total cholesterol (mmol/L) by standardized methods in an automated analyzer (Beckman Coulter-Synchron (Galway, Ireland) in blood samples
Nutritional status | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Albumin (g/dl) by standardized methods in an automated analyzer (Beckman Coulter-Synchron (Galway, Ireland) in blood samples
Nutritional status | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Haemoglobin (g/dl) by standardized methods in an automated analyzer (Beckman Coulter-Synchron (Galway, Ireland) in blood samples
Nutritional status | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Vitamin D (ng/ml) by standardized methods in an automated analyzer (Beckman Coulter-Synchron (Galway, Ireland) in blood samples
Nutritional status | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Vitamin A (ug/dl) by standardized methods in an automated analyzer (Beckman Coulter-Synchron (Galway, Ireland) in blood samples
Nutritional status | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Vitamin E (mg/L) by standardized methods in an automated analyzer (Beckman Coulter-Synchron (Galway, Ireland) in blood samples
Nutritional status | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Carotenoids (ug/dl) by standardized methods in an automated analyzer (Beckman Coulter-Synchron (Galway, Ireland) in blood samples
Cognitive function | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Spanish validated Mini Mental State Examination test (MMSE). The MMSE test various cognitive. The total test score ranges from 0 (impaired) to 30 (normal) (Beaman et al., 2004).
Cognitive function | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  AD8. The AD8 (Alzheimer disease questionnaire) aids in identifying cognitive impairment. This test in combination with the Fototest, significantly increases the diagnosis accuracy of both tests (Carnero Pardo et al., 2012). The optimal cut-off point was 3/4.
Cognitive function | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  TAM test. TAM test (Memory alteration test) provides efficient and valid screening for amnestic Mild Cognitive Impairment and early stage Alzheimer's disease, and discriminates between them. The cut-off score is of 28 points (Rami et al., 2007).
Cognitive function | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Fototest. The Fototest is useful to identify cognitive impairment and dementia in routine clinical practice. (Carnero Pardo et al., 2007). The cut off points are 25/26 for dementia and 28/29 for cognitive impairment.
Brain volume | Visit 1 (week 0), visit 10 (week 36)
  Nuclear Magnetic Resonance (NMR) Total brain volume, hippocampal volume, and volume of white matter hyperintense lesions will be evaluated in a subsample of participants. NMR have allowed important advances in the understanding of age-related brain changes. NMR is a non-invasive instrument that allows the study of the normal aging of individuals at different times of their lives (Barnes et al. 2023).
Cognitive ability assessment | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  BDNF Brain-derived Neutrophic Factor (pg/ml) will be analyzed by Enzyme-linked immunosorbent assay ELISA kit in blood samples
Skeletal muscle strength | Visit 1 (week 0), visit 10 (week 36)
  Isokinetic. Isokinetic test: the evaluation was conducted with an isokinetic dynamometer using a gold standard method (Biodex System 4; Biodex Medical Systems, NewYork, USA) by five repetitions sat two angular velocities (180°s-1, and240°s-1) (Solà et al., 2015). This allows a quantitative evaluation of muscle function through variables such as torque, work and power.
Muscle mass, wasting and turnover | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Muscle mass (skeletal muscle mass (kg)) assessed by Bioimpedance TANITA (MC-780MA; Tanita Corp., Tokyo, Japan).
Muscle mass, wasting and turnover | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Muscle mass (appendicular skeletal muscle mass (kg)) assessed by Bioimpedance TANITA (MC-780MA; Tanita Corp., Tokyo, Japan).
Muscle mass, wasting and turnover | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Muscle mass (skeletal muscle mass index (kg/m2)) assessed by Bioimpedance TANITA (MC-780MA; Tanita Corp., Tokyo, Japan).
Muscle mass, wasting and turnover | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Muscle mass (appedicular skeletal muscle mass index (kg/m2)) assessed by Bioimpedance TANITA (MC-780MA; Tanita Corp., Tokyo, Japan).
Muscle mass, wasting and turnover | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Muscle mass assessed by ultrasound (VINNO 5 (Vinno (Suzhou) Co., Ltd., China)
Muscle mass, wasting and turnover | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Creatine kinase (U/L) assessed by enzymatic assays in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Muscle mass, wasting and turnover | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Cystatin-C (mg/L) assessed by enzymatic assays in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Muscle mass, wasting and turnover | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Serum Myostatin (ng/ml) assessed by commercial ELISA kits (Muscari et al., 2023)
Muscle mass, wasting and turnover | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Serum Follistatin (ng/ml) assessed by commercial ELISA kits (Muscari et al., 2023)
Physical performance | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Gait speed (m/s) assessed by the length of the walking course divided by the time (Ladang et al., 2023).
Signalling pathways in skeletal muscle | Visit 1 (week 0), visit 10 (week 36)
  Muscle gene expression. A muscle biopsy (200-225 mg) will be obtained from a subgroup of volunteers (n=15/group) by trained physicians (Harper et al., 2021). After collection, these samples will be immediately snap frozen in liquid nitrogen and stored at -80°C prior to analysis. To confirm RNA sequencing results obtained in the animal model of age-associated sarcopenia (transcriptomic approach that will be carried out in gastrocnemius skeletal muscle as described in task 5.2), real-time gene expression analysis (qPCR) will be performed, as previously described (Pérez-Matute et al., 2016).
Biological age marker (Aging biomarker) | Visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36)
  Serum N-terminal pro-brain natriuretic peptide (NT-proBNP) (pg/ml) in blood samples (Muscari et al., 2023) is used to diagnose and establish prognosis for heart failure and is a promising biomarker of biological age as it correlates with chronological age and predict life span better than chronological age.
Glucose homeostasis | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  FBG (mmol/L) assessed by standardized methods in an automated analyzer (Beckman Coulter-Synchron, Galway, Ireland) in blood samples
Glucose homeostasis | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Insulin (IU/mL) assessed by standardized methods in an automated analyzer (Beckman Coulter-Synchron, Galway, Ireland) in blood samples
Glucose homeostasis | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  HGBA1c (%) assessed by standardized methods in an automated analyzer (Beckman Coulter-Synchron, Galway, Ireland) in blood samples
Glucose homeostasis | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  HOMA index calculated (Winell et al., 2010) in blood samples
Glucose homeostasis | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  IGF-1 (ng/ml) levels were measured using Human IGF-1 Quantikine ELISA Kit (Pérez-Matute et al., 2022) in blood samples
Lipid profile | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Total cholesterol (mmol/L) in blood samples assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Lipid profile | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  HDLc (mmol/L) in blood samples assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Lipid profile | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  LDLc (mmol/L) in blood samples assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Lipid profile | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  VLDLc (mmol/L) in blood samples assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Lipid profile | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Total TG (mmol/L) in blood samples assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Lipid profile | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  NEFA (mmol/L) in blood samples assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Lipid profile | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  ApoA1 (mg/dL) in blood samples assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Lipid profile | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  ApoB100 (mg/dL) in blood samples assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Lipid profile | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Apo B100/Apo A1 ratio in blood samples assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Lipid profile | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Lp (a) (mg/dL) in blood samples assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Stress Response and Mitochondria | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  GDF15 (pg/mL) Growth differentiating factor 15 is recgonized in mitochondria dysfunction, and as biomarker of aging (Justice et al., 2018) in blood samples
Oxidative markers | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  OxLDL (ug/mL) assessed by commercial ELISA in blood samples
Oxidative markers | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  MetSO/Met (ng/mL) assessed by commercial ELISA in blood samples
Oxidative markers | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  SOD (U/g Hb) 20uL (abcam) in plasma EDTA blood samples assessed by enzymatic assays (Hissin et al., 1976)
Oxidative markers | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  GSHPx (nmol/mL) 50uL (abcam) plasma EDTA blood samples enzymatic assays (Hissin et al., 1976)
Oxidative markers | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  CoQ10 (ug/mL) in blood samples assessed by HPLC
Inflammation markers | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  IL-6 (pg/mL) assessed by immunoturbidimetry on an autoanalyzer (Roche Diagnostics Systems, Madrid, Spain) in blood samples
Inflammation markers | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  hsCRP (mg/L) assessed by immunoturbidimetry on an autoanalyzer (Roche Diagnostics Systems, Madrid, Spain) in blood samples
Inflammation markers | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  TNFRII (pg/mL) assessed by commercial ELISA in blood samples
Inflammation markers | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Adiponectin (ug/mL) assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland) in blood samples
Inflammation markers | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Uric acid (mg/dL) assessed by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland) in blood samples
Vascular parameters | Visit 0, visit 1Visit 0 (week -1), visit 1 (week 0), visit 4 (week 12), visit 7 (week 24), visit 10 (week 36), visit 4, visit 7, visit 10
  Systolic and diastolic blood pressure (SBP and DBP) (mm Hg) and pulse pressure (PP) (mm Hg) assessed by automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain).
Biomarkers of endothelial dysfunction | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  E-selectin (CD62E) (ng/mL) assessed by Commercial ELISA and multi-analyte ELISArray kits as described in our previous work (Catalán et al., 2015) in blood samples
Biomarkers of endothelial dysfunction | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  P-selectin (CD62P) (ng/mL) assessed by Commercial ELISA and multi-analyte ELISArray kits as described in our previous work (Catalán et al., 2015) in blood samples
Biomarkers of endothelial dysfunction | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  ICAM-1 (CD54) (ng/mL) assessed by Commercial ELISA and multi-analyte ELISArray kits as described in our previous work (Catalán et al., 2015) in blood samples
Biomarkers of endothelial dysfunction | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  VCAM-1 (CD106) (ng/mL) assessed by Commercial ELISA and multi-analyte ELISArray kits as described in our previous work (Catalán et al., 2015) in blood samples
Faecal microbial composition | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Metataxonomic profile.
Faecal microbial function | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Microbial functional profile
Faecal metabolome | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  SCFA acetic, butyric, propionic, isobutyric, valeric, isovaleric and caproic acid and phenol colonic metabolites
DNA methylation | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Epigeneitc age. Total genomic DNA will be extracted from saliva samples using the Norgen Saliva DNA Isolation Kit.
Gut permeability determined on plasma | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Zonulin (ng/mL). Human zonulin levels will be quantified using an ELISA kit (Cusabio® Technology Llc, Houston, TX, USA)
Biomarkers of wine intake compliance | Visit 1 (week 0), visit 7 (week 24), visit 10 (week 36)
  Quantification of urine phenol metabolites in human elderly

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà Alberich, Professor, Principal Investigator — Universitat Rovira i Virgili, Facultat de Medicina i Ciències de la Salut, NFOC-Salut group, 43201 Reus, Spain Institut Investigació Sanitària Pere i Virgili (ISPV), 43204, Reus, Spain Hospital Universitari Sant Joan de Reus, 43204, Reus, Spain; Anna Pedret Figuerola, Dr., Principal Investigator — Universitat Rovira i Virgili, Facultat de Medicina i Ciències de la Salut, NFOC-Salut group, 43201 Reus, Spain
Locations (1):
- Universitat Rovira i Virgili, Facultat de Medicina i Ciències de la Salut, Functional Nutrition, Oxidation, and Cardiovascular Diseases Group (NFOC-Salut), Reus, Spain, Spain

IPD SHARING:
Plan to Share IPD: No